CLINICAL TRIAL: NCT01719848
Title: Evaluation of Clinical Airway Assessments for Predicting Difficult Laryngoscopy Using a Gray Zone Approach
Brief Title: Evaluation of Clinical Airway Assessments With a Gray Zone Approach
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, assistant professor, Samsung Medical Center
Other Study IDs: 2012-05-079-001
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Difficult Laryngoscopy
Keywords: Physical examinations, Percentage of glottic opening(POGO)
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preoperative airway examination: patients undergoing general anesthesia for any surgery
  Interventions: Other: Measurements of parameters related with physical examinations for difficult airway prediction

INTERVENTIONS:
Other: Measurements of parameters related with physical examinations for difficult airway prediction

SUMMARY:
Failure of advanced airway security has been reported that it could lead lethal complication such as brain hypoxic damage. There have been controversial reports for the airway assessment tests which can predict difficult laryngoscopy. Therefore, we evaluated diagnostic validity of pre-existing airway assessment tests and scoring system using a gray zone approach in patients undergoing general anesthesia required endotracheal intubation.

DETAILED DESCRIPTION:
POGO(percentage of glottic opening)will be evaluated by an attachable fiberoptic scope (AV scope. CAREtec CO.Ltd, Kangwon-Do, South Korea)

ELIGIBILITY:
Inclusion Criteria:

* 20 to 80 years old patients undergoing general anesthesia for any operation.

Exclusion Criteria:

* previous difficult airway history
* upper airway obstruction disease
* congenital disorders that are known to relate with difficult airway
* neurologic symptom associated with neck extension
* emergent operation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia for any surgery at Samsung medical center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percentage of glottic opening (POGO) | During laryngoscopy manipulation for endotracheal intubation (average 3min after muscle relaxant is delivered)
  POGO image will be captured using attachable fiberoptic scope.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Derived] Min JJ, Kim G, Kim E, Lee JH. The diagnostic validity of clinical airway assessments for predicting difficult laryngoscopy using a grey zone approach. J Int Med Res. 2016 Aug;44(4):893-904. doi: 10.1177/0300060516642647. Epub 2016 Jun 6. PMID 27268499